CLINICAL TRIAL: NCT06659783
Title: The First Acute Upper Gastrointestinal Bleeding (AUGIB) Audit in the Greater Bay Area (GBA) of China
Acronym: AUGIB Audit
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, MD, Professor, Chinese University of Hong Kong
Other Study IDs: AUGIB Audit GBA
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: AUGIB; Gastrointestinal Bleeding
Keywords: AUGIB; audit; Greater Bay Area; GBA; epidemiology
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unselected acute UGIB adult patients admitted with overt signs of AUGIB or in-bleeder: 40 hospitals receiving emergency admissions in the Guangdong-Hong Kong-Macao area in China are invited to participate in this study. Unselected acute UGIB adult patients (≥18 years old) admitted within a 2-month period in the second quarter of 2025 are identified. These patients are newly admitted patients from both the emergency department and clinics with overt signs of AUGIB, as well as patients who develop bleeding while hospitalized for other reasons.

SUMMARY:
Investigators aim to conduct a large-scale, prospective cohort study in the Greater Bay Area of South China. Investigators aim to identify consecutive patients with AUGIB in the area over a 2-month period in the second quarter of 2025.

This study covers the Guangdong-Hong Kong-Macao Greater Bay Area (GBA) as well as the western, eastern, and northern regions of Guangdong Province. It comprises of 2 Special Administrative Regions of Hong Kong and Macao and 21 municipalities in Guangdong Province (Guangzhou, Shenzhen, Foshan, Dongguan, Zhongshan, Zhuhai, Jiangmen, Zhaoqing, Huizhou, Shantou, Chaozhou, Jieyang, Shanwei, Zhanjiang, Maoming, Yangjiang, Yunfu, Shaoguan, Qingyuan, Meizhou, Heyuan). The total population of the Guangdong-Hong Kong-Macao area is estimated to be 135.24 million. Investigators aim to understand the current epidemiology of AUGIB in South China by collecting patient characteristics, the care model and management strategies including the use of endoscopy, interventional radiology and surgery, and the associated mortality.

The goal is to identify areas for improving patients' outcomes and to reduce mortality. The audit also provides a reference standard for future audits and a comparison to a minimal international standard.

Acute Upper gastrointestinal bleeding (AUGIB) remains a common medical emergency. Although the annual incidence of AUGIB has decreased from approximately 100 per 100,000 adults in the 1990s to 61-78 per 100,000 persons in 2009-2012, the 30-day mortality rate remains as high as 11%. The overall etiology and epidemiology of acute UGIB have undergone significant changes. The widespread eradication of H. pylori, the use of safer non-steroidal anti-inflammatory drugs (NSAIDs), and the use of proton pump inhibitors (PPIs) have reduced the incidence of bleeding peptic ulcers. The increasing prevalence of alcohol-related liver disease, common usage of anticoagulant or antiplatelet therapy, and an aging population (with associated co-morbidities) often worsen the prognosis. Overall, in the management of patients with AUGIB, the diagnostic and treatment methods such as endoscopic hemostasis have improved. This together with better access to both high-dependency care and interventional radiology can all contribute to better patient outcome in acute UGIB.

Epidemiologic studies in acute upper gastrointestinal hemorrhage from Asia mostly come from hospital-based studies with limited number of cases. These studies are largely retrospective in their nature. In China, there is a lack of population-based studies on AUGIB. There are also uncertainties in how these patients are managed especially over adoption of risk stratification tools, timely provision of care, the use of endoscopic hemostatic treatment, the use of drugs and red cell transfusion, and interventional radiology.

To understand the current epidemiology of AUGIB in the GBA, investigators aim to conduct a large-scale, prospective cohort study in the Greater Bay Area of South China. In this audit, Investigators identify patients with AUGIB admitted to participating hospitals and collect their demographic data, clinical presentation, management and outcomes The goal is to identify areas of opportunities in reducing mortality and improving patient outcomes.

This is a population based, unselected multicentre, prospective survey. Consecutive patients who present with signs of AUGIB, aged >18, admitted to the participating hospitals from August 1, 2024, to September 30, 2024, are identified. These patients include those admitted through the emergency department, and clinics, and patients who develop bleeding while being hospitalized for other reasons.

DETAILED DESCRIPTION:
Up to forty hospitals receiving emergency admissions in the Guangdong-Hong Kong-Macao area in China are invited to participate in this study. Unselected acute UGIB adult patients (≥18 years old) admitted within a 2-month period in the second quarter of 2025 are identified. These patients are newly admitted patients from both the emergency department and clinics with overt signs of AUGIB, as well as patients who develop bleeding while hospitalized for other reasons At each center a "lead" consultant is designated to represent the hospital on the project. Lead PI and designated research staff identify cases by screening admission records to accident and emergency department and the admission wards, records in the endoscopy centre, interventional radiology suites and operating theater, and through direct communication with admitting staff at respective clinical area. To ensure completeness of case ascertainment, an audit coordinator will cross check data entry against hospital admission, discharge records including records of the deceased. For each identified, the site PI and designated research staff will extract relevant data to complete an audit questionnaire and enter the data into a secure web-based Case Report Form, which can only be accessed using a unique hospital identifier and password. All records are anonymized. The following information is being collected. A central audit coordinator checks at weekly interval completeness of questionnaire entry and communicate with site research staff for clarification.

Information extracted included demographics, clinical history (such as admission date, time, clinical areas , referral pattern, past medical history, signs and symptoms at presentation, observations at time of presentation for the clinical episode), laboratory tests, medications, interventions and clinical outcomes

Acute upper gastrointestinal bleeding is deﬁned as the passage of melaena and/or ﬁrm clinical evidence and laboratory support for acute blood loss from the upper gastrointestinal (UGI) tract.

This is an observational study. All patients are managed per each center's standard of care. Therefore, no extra intervention is administered and thus there would be no adverse effects expected from the present study. In each enrolled centre, a "lead" consultant together with designated research staff including at least a medical doctor and an audit coordinator will make sure all data are collected correctly and faithfully. The lead investigator of the study will be in direct contact with each centre for any problem related to the study.

This is an observational study. All patients are managed and followed up per each center's standard of care. Therefore, no extra intervention is administered.

Data are presented as percentages with numerator/denominator and as summary statistics of median and inter-quartile ranges (IQR) or mean (standard deviation) as appropriate. Binary regression methods are used to calculate risk ratios and 95% confidence intervals to assess the association of clinical factors with outcomes (inpatient mortality, re-bleeding, red blood cell transfusion). Risk ratios for the type of admission, co-morbidities, and alcohol abuse were computed after adjusting for patient age, which was categorized into quintiles.

At each center a "lead" consultant is designated to represent the hospital on the project. Lead PI and designated research staff identify cases by screening admission records to accident and emergency department and the admission wards, records in the endoscopy centre, interventional radiology suites and operating theater, and through direct communication with admitting staff at respective clinical area. To ensure completeness of case ascertainment, an audit coordinator will cross check data entry against hospital admission, discharge records including records of the deceased. For each identified, the site PI and designated research staff will extract relevant data to complete an audit questionnaire and enter the data into a secure web-based Case Report Form, which can only be accessed using a unique hospital identifier and password. All records are anonymized. The following information is being collected. A central audit coordinator checks at weekly interval completeness of questionnaire entry and communicate with site research staff for clarification.

Information extracted included demographics, clinical history (such as admission date, time, clinical areas , referral pattern, past medical history, signs and symptoms at presentation, observations at time of presentation for the clinical episode), laboratory tests, medications, interventions and clinical outcomes

Acute upper gastrointestinal bleeding is deﬁned as the passage of melaena and/or ﬁrm clinical evidence and laboratory support for acute blood loss from the upper gastrointestinal (UGI) tract.

This is an observational study. All patients are managed per each center's standard of care. Therefore, no extra intervention is administered and thus there would be no adverse effects expected from the present study. In each enrolled centre, a "lead" consultant together with designated research staff including at least a medical doctor and an audit coordinator will make sure all data are collected correctly and faithfully. The lead investigator of the study will be in direct contact with each centre for any problem related to the study.

This is an observational study. All patients are managed and followed up per each center's standard of care. Therefore, no extra intervention is administered.

Data are presented as percentages with numerator/denominator and as summary statistics of median and inter-quartile ranges (IQR) or mean (standard deviation) as appropriate. Binary regression methods are used to calculate risk ratios and 95% confidence intervals to assess the association of clinical factors with outcomes (inpatient mortality, re-bleeding, red blood cell transfusion). Risk ratios for the type of admission, co-morbidities, and alcohol abuse were computed after adjusting for patient age, which was categorized into quintiles.

For each included case, the audit coordinator will extract relevant data to complete the audit questionnaires and enter the data into a secure web-based Case Report Form, which can only be accessed using a unique hospital identifier and password. Data will be electronically exported from the website into SPSS. Any duplicate cases will be identified and removed from the dataset prior to analysis. Dates (e.g., date of admission, date of endoscopy, date of discharge) will be verified, and free-text comments regarding presentation and diagnoses were reclassified where possible. Clinical leads will be contacted for clarification when necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients would be included in the study if they are aged 18 years or older and have clinical evidence of AUGIB on admission, or clinical evidence of AUGIB while as an inpatient for any other reason. We also include patients with hematochezia as some patients with brisk AUGIB can present rectal bleeding

Exclusion Criteria:

* Patients younger than 18 years old.
* Patients presenting with iron deﬁciency anemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 hospitals receiving emergency admissions in the Guangdong-Hong Kong-Macao area in China are invited to participate in this study. Unselected acute UGIB adult patients (≥18 years old) admitted within a 2-month period in the second quarter of 2025. These patients are newly admitted patients from both the emergency department and clinics with overt signs of AUGIB, as well as patients who develop bleeding while hospitalized for other reasons.
Sampling Method: Non-Probability Sample
Enrollment: 4534 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-01-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  Mortality of all causes

CONTACTS AND LOCATIONS:
Overall Officials: Side Liu, PhD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (40):
- China (39):
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Dongguan Songshan Lake Tungwah Hospital, Dongguan, Guangdong
  - Donghua Hospital, Dongguan, Dongguan, Guangdong
  - Houjie Hospital of Dongguan, Dongguan, Guangdong
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - Guangzhou Red Cross Hospital, Guangzhou, Guangdong
  - Huadu District People's Hospital, Guangzhou, Guangdong
  - The Affiliated Panyu Central Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University (Guangzhou Overseas Chinese Hospital), Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangzhou Eighth People's Hospital, Guangzhou Medical University, Guangzhou, Guangdong
  - Southern Medical University Zhujiang Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Huizhou First People's Hospital, Huizhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Wuyi Hospital of Traditional Chinese Medicine, Jiangmen, Guangdong
  - Huazhong University of Science and Technology Union Hospital (Nanshan Hospital), Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Longgang Central Hospital of Shenzhen, Shenzhen, Guangdong
  - Longgang District People's Hospital, Shenzhen (The Second Affiliated Hospital of The Chinese University of Hong Kong, Shenzhen), Shenzhen, Guangdong
  - Longhua New District People's Hospital, Shenzhen, Shenzhen, Guangdong
  - Southern Medical University Shenzhen Hospital, Shenzhen, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University Zhaoqing Hospital, Zhaoqing, Guangdong
  - Zhaoqing First People's Hospital, Zhaoqing, Guangdong
  - Huoju Development District Hospital, Zhongshan, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - Foshan First People's Hospital, Zhuhai, Guangdong
  - Foshan Second People's Hospital, Zhuhai, Guangdong
  - Southern Medical University Shunde Hospital, Zhuhai, Guangdong
  - The Fifth Affiliated Hospital of Zunyi Medical University, Zhuhai - Foshan City (3 Centers), Zhuhai, Guangdong
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - Guangzhou First People's Hospital, Guangdong, guangzhou
  - Kiang Wu Hospital, Macao, Macao
- Chinese University of Hong Kong, Shatin, Hong Kong SAR, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Laine L, Spiegel B, Rostom A, Moayyedi P, Kuipers EJ, Bardou M, Sung J, Barkun AN. Methodology for randomized trials of patients with nonvariceal upper gastrointestinal bleeding: recommendations from an international consensus conference. Am J Gastroenterol. 2010 Mar;105(3):540-50. doi: 10.1038/ajg.2009.702. Epub 2009 Dec 22. PMID 20029415
- [Background] Siau K, Hearnshaw S, Stanley AJ, Estcourt L, Rasheed A, Walden A, Thoufeeq M, Donnelly M, Drummond R, Veitch AM, Ishaq S, Morris AJ. British Society of Gastroenterology (BSG)-led multisociety consensus care bundle for the early clinical management of acute upper gastrointestinal bleeding. Frontline Gastroenterol. 2020 Mar 27;11(4):311-323. doi: 10.1136/flgastro-2019-101395. eCollection 2020. PMID 32582423
- [Background] Hearnshaw SA, Logan RF, Lowe D, Travis SP, Murphy MF, Palmer KR. Acute upper gastrointestinal bleeding in the UK: patient characteristics, diagnoses and outcomes in the 2007 UK audit. Gut. 2011 Oct;60(10):1327-35. doi: 10.1136/gut.2010.228437. Epub 2011 Apr 13. PMID 21490373
- [Background] Barkun AN, Almadi M, Kuipers EJ, Laine L, Sung J, Tse F, Leontiadis GI, Abraham NS, Calvet X, Chan FKL, Douketis J, Enns R, Gralnek IM, Jairath V, Jensen D, Lau J, Lip GYH, Loffroy R, Maluf-Filho F, Meltzer AC, Reddy N, Saltzman JR, Marshall JK, Bardou M. Management of Nonvariceal Upper Gastrointestinal Bleeding: Guideline Recommendations From the International Consensus Group. Ann Intern Med. 2019 Dec 3;171(11):805-822. doi: 10.7326/M19-1795. Epub 2019 Oct 22. PMID 31634917
- [Background] Wuerth BA, Rockey DC. Changing Epidemiology of Upper Gastrointestinal Hemorrhage in the Last Decade: A Nationwide Analysis. Dig Dis Sci. 2018 May;63(5):1286-1293. doi: 10.1007/s10620-017-4882-6. Epub 2017 Dec 27. PMID 29282637
- [Background] Laine L, Yang H, Chang SC, Datto C. Trends for incidence of hospitalization and death due to GI complications in the United States from 2001 to 2009. Am J Gastroenterol. 2012 Aug;107(8):1190-5; quiz 1196. doi: 10.1038/ajg.2012.168. Epub 2012 Jun 12. PMID 22688850
- [Background] Abougergi MS, Travis AC, Saltzman JR. The in-hospital mortality rate for upper GI hemorrhage has decreased over 2 decades in the United States: a nationwide analysis. Gastrointest Endosc. 2015 Apr;81(4):882-8.e1. doi: 10.1016/j.gie.2014.09.027. Epub 2014 Dec 5. PMID 25484324
- [Background] Sung JJ, Chiu PW, Chan FKL, Lau JY, Goh KL, Ho LH, Jung HY, Sollano JD, Gotoda T, Reddy N, Singh R, Sugano K, Wu KC, Wu CY, Bjorkman DJ, Jensen DM, Kuipers EJ, Lanas A. Asia-Pacific working group consensus on non-variceal upper gastrointestinal bleeding: an update 2018. Gut. 2018 Oct;67(10):1757-1768. doi: 10.1136/gutjnl-2018-316276. Epub 2018 Apr 24. PMID 29691276
- [Background] Kwan I, Bunn F, Chinnock P, Roberts I. Timing and volume of fluid administration for patients with bleeding. Cochrane Database Syst Rev. 2014 Mar 5;2014(3):CD002245. doi: 10.1002/14651858.CD002245.pub2. PMID 24599652
- [Background] Rosenstock SJ, Moller MH, Larsson H, Johnsen SP, Madsen AH, Bendix J, Adamsen S, Jensen AG, Zimmermann-Nielsen E, Nielsen AS, Kallehave F, Oxholm D, Skarbye M, Jolving LR, Jorgensen HS, Schaffalitzky de Muckadell OB, Thomsen RW. Improving quality of care in peptic ulcer bleeding: nationwide cohort study of 13,498 consecutive patients in the Danish Clinical Register of Emergency Surgery. Am J Gastroenterol. 2013 Sep;108(9):1449-57. doi: 10.1038/ajg.2013.162. Epub 2013 Jun 4. PMID 23732464